CLINICAL TRIAL: NCT04600700
Title: Real-time Continuous Predictive Analytics Algorithm to Optimize Weaning of Inotropic Agents in Post-operative Pediatric Surgical Cardiac Patients
Brief Title: Use of a Predictive Analytics Algorithm to Optimize Weaning of Inotropes Following Pediatric Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joshua Salvin, Cardiac Intensive Care Physician, Boston Children's Hospital
Other Study IDs: P00036870; R44HL117340 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Congenital Heart Disease
Keywords: cardiac surgery; congenital heart disease; critical care; pediatrics
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CDSS weaning group: This group will be exposed to the CDSS to inform inotrope weaning
  Interventions: Device: Clinical Decision support system (CDSS) for inotrope weaning

INTERVENTIONS:
Device: Clinical Decision support system (CDSS) for inotrope weaning — A Clinical Decision Support System informed by 6-hour rolling average IDO2, will be utilized during the intervention phase of the study. The CDSS tool will be introduced in a stepped-wedge pattern. Randomization will occur by center, with time of introduction being staggered, with each center ultimately receiving the CDSS intervention. Teams in the CICU make rounds twice per day. During each of the rounds (AM and PM), the team will refer to the CDSS and the 6-hour average IDO2 (as reported on the T3 platform at the bedside computer). The clinical team will consider the CDSS in decision making around inotrope weans. If the decision is made to not utilize IDO2, the bedside clinician will complete a brief survey with rationale.

SUMMARY:
The objective of this study is to determine the effectiveness of a real time continuous risk analytics algorithm in the successful de-escalation of vasoactive and inotropic support in pediatric patients following cardiac surgery.

DETAILED DESCRIPTION:
IDO2 utilizes high fidelity continuous and intermittent patient data to feed a Bayesian model which predicts the risk of inadequate tissue oxygen delivery. This index (the IDO2) is FDA 510k cleared for pediatric patients 2 kg up to 12 years of age to continuously report the risk for inadequate tissue oxygen delivery (defined as a mixed venous oxygen saturation less than 40%). The index is continuously displayed in graphical form at the bedside. Clinical decision support systems (CDSS) such as IDO2 may inform inform the clinician when it is appropriate to de-escalate care on a critically ill. Appropriate de-escalation plays a role in the safe, efficient utilization of resources in the CICU, and may reduce duration intervals of care such as duration of support with vasoactive and inotropic drugs, mechanical ventilation and length of stay. In support of this hypothesis, the investigators for this proposed study have recently completed a retrospective, multi-center analysis of 2,556 patient encounters demonstrating that elevated IDO2 during a wean off inotropic agents is associated with weaning failure. When compared to conventional markers of cardiac output, 6-hour average IDO2 was superior to lactate elevation, fall in base deficit, and fall in urine output in discriminating inotrope weaning success from failure. Additionally, for those patients who failed inotrope wean, rescue with re-starting an inotrope was associated with a concomitant fall in IDO2. This analysis supports an underlying hypothesis that IDO2 reflects underlying patient stability, and the rescue of deteriorating physiology leads to an improved physiologic state, and hence a lower IDO2.7 Data suggest that simple CDSS which prompt discussion about management decisions, such as those made during daily ICU rounds, may improve outcomes. These CDSS are often in the form of checklists and apply to usual or standardized practices. These simplified mechanisms may not apply to the more dynamic clinical situations in which specific and intensively monitored patient populations can demonstrate variable response to drugs and recovery. In these circumstances, a CDSS utilizing a 6-hour rolling average value of IDO2, in which the physiologic response to decisions is demonstrated continuously, may inform a more rapid more efficient and safe de-escalation of vasoactive and inotropic drugs when implemented on each of the twice daily clinical work rounds in the CICU.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants aged 1-365 days
* weight greater than 3kg
* Gestational age greater than 36 weeks
* admitted to the cardiovascular intensive care uni following biventricular repairs of congenital heart disease
* high risk for hemodynamic instability (ie started on inotropes - milrinone, epinephrine, norepinephrine, dopamine, vasopressin) in operating room or within 6 hours cardiopulmonary bypass cessation.

Exclusion Criteria:

* Patients undergoing palliation of single ventricle heart disease
* surgical cases not requiring cardiopulmonary bypass
* cases not requiring vasoactive or inotropic support
* patients requiring extracorporeal membrane oxygenation (ECMO) in the perioperative period (either out of the operating room, or in the ICU prior to weaning off inotropic support)
* patients who died prior to weaning off inotropic support

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates and infants with congenital heart disease following cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Hours of inotropic support | 12/31/21
  Hours of inotropic support

SECONDARY OUTCOMES:
Hours of mechanical ventilation | 12/31/21
  Hours of mechanical ventilation
Days in the Cardiac Intensive Care Unit (CICU) | 12/31/21
  Number of days in the CICU
Number of central line days | 12/31/21
  Number of days with a central catheter
Rate of nosocomial infection | 12/31/21
  The rate per patient day of nosocomial infection
adherence to Clinical Decision Support System (CDSS) | 12/31/21
  Number of deviations from the protocol
hospital cost | 12/31/21
  Hospital charges in US dollars

CONTACTS AND LOCATIONS:
Overall Officials: Joshua W Salvin, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gazit AZ, Futterman C, Baronov D, Tomczak A, Goldsmith MP, Talisa VB, Nadkarni VM, Laussen PC, Salvin JW. Risk Analytics Clinical Decision Support Decreases Duration of Vasoactive Infusions Following Pediatric Cardiac Surgery: A Multicenter Before and After Clinical Trial. Crit Care Med. 2025 Jul 1;53(7):e1355-e1364. doi: 10.1097/CCM.0000000000006682. Epub 2025 Apr 29. PMID 40298483